CLINICAL TRIAL: NCT01477229
Title: Quality of Life in RECTal Cancer - A Study Within the Scandinavian Surgical Outcomes Research Group
Brief Title: Quality of Life in RECTal Cancer - a Prospective Multicenter Cohort Study
Acronym: QoLiRECT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Swedish Cancer Foundation (Other); The Swedish Society of Medicine (Other); Assar Gabrielsson Foundation (Unknown)
Responsible Party: Principal Investigator, Eva Angenete, M.D., Ph.D, Sahlgrenska University Hospital
Other Study IDs: QoLiRECT
Record Dates: First submitted 2011-11-15; First posted 2011-11-22 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Rectal Cancer; Quality of Life; Surgery
Keywords: Rectal cancer; Quality of Life; Abdominoperineal Resection; Anterior Resection; Palliative cancer treatment; Radio chemotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Abdominoperineal resection: Patients with low rectal cancers
- Anterior resection: Patients where it is possible to perform an anterior resection
- Preoperative chemo-radiation treatment: Patients with locally advanced rectal cancer
- Palliative treatment: Patients with systemic disease

SUMMARY:
Rectal cancer is a common type of cancer occuring more frequently in men but also common in women. Almost 60% of the patients survive 5-years and the treatment has been continuously developed in the last three decades. The aim of the QoLiRECT study is to increase the knowledge about symptoms, functional impairments, quality of life (QoL) and psychological and socioeconomic burden in an unselected population of rectal cancer patients.

DETAILED DESCRIPTION:
Rectal cancer is more frequent in men than in women and is relatively uncommon before the age of 50. The prognosis for rectal cancer has improved over the last decades2. Almost 60% of all patients survive more than five years, and because of advances in early detection and treatment, this number is expected to increase in the future1. Treatment of rectal cancer varies depending on the stage of the disease at diagnosis. For some patients, operation is the only treatment. For others, surgery is combined with radiotherapy, chemotherapy or both. The two most common operative procedures are the sphincter-preserving anterior resection (AR) and the abdominoperineal resection (APR) - the latter results in a permanent colostomy. Patients with generalised disease at diagnosis receive palliative treatment, which may include chemotherapy and radiotherapy as well as surgery.

Rectal cancer comes with a high risk of local recurrence, i.e. return of the tumour within the pelvis after a presumed curative resection. Local recurrence is difficult to treat and often very painful and distressing for the patient. Some local recurrences will be candidates for second line surgery, as is also true for some distant metastases.

The aim of the QoLiRECT study is to increase the knowledge about symptoms, functional impairments, quality of life (QoL) and psychological and socioeconomic burden in an unselected population of rectal cancer patients. Symptoms such as incontinence, pain, fatigue and impaired sexual function3 are common with this disease. Bodily changes, caused by the treatment or the disease itself, may lead to functional impairments and psychological, social, emotional and economical restraints. Conventional outcome measures such as morbidity and survival reveal little about these things.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting at the participating hospitals with newly diagnosed rectal cancer, regardless of stage at diagnosis and plans for treatment, will be eligible for inclusion.

Exclusion Criteria:

* Age below 18 years at diagnosis.
* No informed consent received or withdrawal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting at the participating hospitals (both University Hospitals and Community Hospitals) with newly diagnosed rectal cancer, regardless of stage at diagnosis and plans for treatment, will be eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To describe QoL, symptoms and functional impairments in an unselected population of rectal cancer patients | At diagnosis
  It will be evaluated at diagnosis, , i.e. at presentation of a plan for the treatment, at 12 months after start of the treatment, regardless of which, at 24 months after start of the treatment and at 60 months after start of the treatment

SECONDARY OUTCOMES:
To explore potential differences in QoL, symptoms and functional impairments between subgroups of the population | At diagnosis
  and at 12 months, 36 months and 60 monts after diagnosis
To identify symptoms and functional impairments and other risk factors that have great impact on QoL | At diagnosis
  will also be assessed at 12 months after start of the treatment, regardless of which, at 24 months after start of the treatment and at 60 months after start of the treatment
To identify patient and environmental factors with an impact on QoL | At diagnosis
  and at 12 months after start of the treatment, regardless of which, at 24 months after start of the treatment and at 60 months after start of the treatment
To analyse how clinical factors like oncologic result of operation, morbidity, recurrence and survival influence QoL | At 12 months after start of the treatment
  This will be analyzed regardless of which, at 24 months after start of the treatment and at 60 months after start of the treatment
To initiate interventional studies when appropriate | 12 months
  May be another time frame than the one registered. Depends on results from the QoL questionnaire
To generate basic descriptive data of the rectal cancer patient population: demography, socioeconomic data, disease stage at diagnosis, fashion of treatment, recurrence, survival | At diagnosis
To analyse health economy aspects of QoL and morbidity in the patient population | At diagnosis
  and at 12 months after start of the treatment, regardless of which, at 24 months after start of the treatment and at 60 months after start of the treatment
To explore the presence and impact of intrusive thoughts on QoL | At 12 months
  May be analyzed both at 24 and 60 months as well
QoL in an unselected population of rectal cancer patients | at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, M.D., Ph.D., Principal Investigator — SSORG - Scandinavian Surgical Outcomes Research Group and Sahlgrenska University Hospital in collaboration with Sahlgrenska Academy at University of Gothenburg
Locations (1):
- Scandinavian Surgical Outcomes Research Group, SSORG, Göteborg, Gothenburg, Sweden

REFERENCES:
- [Derived] Bjorklund Sand L, Larsson C, Gronkvist R, Haglind E, Angenete E. Persistent Sitting and Walking Difficulties After Abdominoperineal Excision and Anterior Resection: Results From the Quality of Life in Rectal Cancer Study. Dis Colon Rectum. 2025 Jun 1;68(6):704-712. doi: 10.1097/DCR.0000000000003710. Epub 2025 Mar 14. PMID 40085057
- [Derived] Ehrencrona C, Li Y, Angenete E, Haglind E, Franzen S, Grimby-Ekman A, Bock D. Do beta-blockers reduce negative intrusive thoughts and anxiety in cancer survivors? - An emulated trial. BMC Cancer. 2024 Apr 11;24(1):447. doi: 10.1186/s12885-024-12236-3. PMID 38605350
- [Derived] Asplund D, Heath J, Gonzalez E, Ekelund J, Rosenberg J, Haglind E, Angenete E. Self-reported quality of life and functional outcome in patients with rectal cancer--QoLiRECT. Dan Med J. 2014 May;61(5):A4841. PMID 24814743